CLINICAL TRIAL: NCT00576836
Title: Dose Study of Thymus Transplantation in DiGeorge Anomaly, IND 9836, #932.1
Brief Title: Thymus Transplantation Dose in DiGeorge #932
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016144; FDA-FD-R-002606 (Other Grant/Funding Number: FDA OOPD); 2R01AI047040-11A2 (NIH); R56 Bridge R01AI4704011A1 (Other Grant/Funding Number: NIH American Recovery and Reinvestment Act (ARRA) of 2009); 5K12HD043494-09 (NIH); R01AI054843 (NIH); R01AI047040 (NIH); 3R56AI047040-11A1S1 (NIH); 932 (Other: Duke)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: DiGeorge Anomaly; DiGeorge Syndrome; Complete DiGeorge Anomaly; Complete DiGeorge Syndrome
Keywords: Thymus Transplantation; DiGeorge Syndrome; DiGeorge Anomaly; Athymia; Parathyroid Transplantation; Hypocalcemia; Hypoparathyroidism; Low T cell numbers; Immunoreconstitution; Immunodeficiency; Complete DiGeorge; Complete DiGeorge Anomaly; Typical DiGeorge; Cultured Thymus Tissue Implantation (CTTI)
MeSH Terms: conditions — DiGeorge Syndrome; Thymic aplasia; Hypocalcemia; Hypoparathyroidism; Immunologic Deficiency Syndromes | interventions — Transplantation; Thymus Extracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cultured Thymus Tissue Implantation w Parathyroid Transplant (Experimental): Cultured Thymus Tissue Implantation With Parathyroid Tissue Transplantation. Subjects who were enrolled in this arm underwent cultured thymus tissue implantation with parathyroid transplantation, if eligible.
  No specific dose was assigned. The thymus tissue dose was the number of grams of cultured thymus tissue divided by the weight of the recipient in kg or per square meter of body surface area of the recipient.
  There was a one time administration of the cultured thymus tissue and parathyroid tissue.
  Interventions: Other: Cultured Thymus Tissue Implantation with Parathyroid Transplantation
- Cultured Thymus Tissue Implantation (Experimental): Cultured Thymus Tissue Implantation. Subjects who were enrolled in this arm underwent cultured thymus tissue implantation (CTTI) only.
  No specific dose was assigned. The thymus tissue dose was the number of grams of cultured thymus tissue divided by the weight of the recipient in kg or per square meter of body surface area of the recipient.
  There was a one time administration of the cultured thymus tissue.
  .
  Interventions: Biological: Cultured Thymus Tissue Implantation (CTTI)

INTERVENTIONS:
Biological: Cultured Thymus Tissue Implantation (CTTI) — Thymus tissue (from unrelated donor), thymus donor, and thymus donor's birth mother screened for safety. CTTI was done under general anesthesia. Cultured thymus tissue was implanted into quadriceps. Thymus dose at least 4grams/m2 body surface area (0.2 grams/kg body weight) and not >18 grams/m2 body surface area (1.0 grams/kg body weight). At time of CTTI, skin biopsy was obtained to look for preexisting T cells. 2-3 months post-CTTI allograft biopsy was done to evaluate for thymopoiesis & graft rejection. At time of biopsy, skin biopsy done to look for T cell clonal populations. (Allograft biopsy not done if subject medically unstable.) Post-CTTI, subjects followed by immune evaluations, using blood samples.
  Other Names: Thymus Tissue for Transplantation; CTTI
  Arms: Cultured Thymus Tissue Implantation
Other: Cultured Thymus Tissue Implantation with Parathyroid Transplantation — Parental parathyroid donors screened for eligibility and safety. If both parents meet eligibility criteria, the parathyroid will be harvested from parent who shares the most Human Leukocyte Antigens (HLA) alleles with thymus donor. Parathyroid harvest & transplant preferably done at same time as CTTI. (If parathyroid transplant cannot be done at same time, then it is done within 3-8 weeks of CTTI.) Parathyroid harvest done under general anesthesia. One parathyroid gland is minced & placed in quadriceps muscle; there is no dose in mg. No biopsy done of the parathyroid. Parathyroid donors are monitored as outpatients until recipients' discharge. Recipients' calcium and PTH levels are monitored indefinitely.
  Other Names: Thymus and Parathyroid Transplant; CTTI and Parathyroid Transplant
  Arms: Cultured Thymus Tissue Implantation w Parathyroid Transplant

SUMMARY:
One purpose of this study is to determine whether the amount of cultured thymus tissue implanted into DiGeorge anomaly infants has any effect on the immune outcome. Another purpose of this study is to determine whether parental parathyroid transplantation (in addition to cultured thymus tissue implantation (CTTI) can help both the immune and the calcium problems in DiGeorge infants with hypocalcemia. [Funding Source - FDA Office of Orphan Products Development (OOPD)]

DETAILED DESCRIPTION:
DiGeorge anomaly is a congenital disorder in which infants are born with defects of the thymus, heart, and parathyroid gland. Complete DiGeorge Anomaly is usually fatal within the first two years of life. This trial evaluates the role of cultured thymus tissue dose in cultured thymus tissue implantation (CTTI) in complete (typical) DiGeorge anomaly infants, and continues safety assessments.

DiGeorge infants who have successful CTTIs but remain with hypoparathyroidism must go to the clinic for frequent calcium levels and to the hospital for calcium infusions; these infants are at risk for seizures from low calcium. Approximately ½ of infants with profound hypoparathyroidism will develop nephrocalcinosis. This protocol had a parental parathyroid transplant arm for complete DiGeorge infants with athymia and profound hypoparathyroidism.

ELIGIBILITY:
Thymus Transplant Inclusion Criteria:

* A parent or guardian of the DGS subject signed the consent form.
* Medical screening was completed.
* For a diagnosis of DGS, the subject had to have one of the following:

  * Congenital heart disease;
  * Hypocalcemia requiring replacement;
  * 22q11.2 hemizygosity or 10p13 hemizygosity;
  * CHARGE association or CHD7 mutation;
  * A subject with abnormal ears whose mother had diabetes (type I, type II, or gestational).
* To meet the criteria of typical complete DiGeorge Anomaly (cDGA), the subject had to have either:

  * Circulating CD3+ T cell count by flow cytometry < 50/mm3 OR
  * Circulating CD3+ T cells that were also positive for Cluster of Differentiation 45RA (CD45RA)+ CD62L+ and were < 50/mm3 or less than 5% of total T cells.

Thymus Transplant Exclusion Criteria:

* Had heart surgery less than 4 weeks prior to projected implant date;
* Heart surgery anticipated within 3 months after the proposed time of implantation;
* Present or past lymphadenopathy;
* Rash associated with T cell infiltration of the dermis and epidermis;
* Rejection by the surgeon or anesthesiologist as surgical candidate;
* Lack of sufficient muscle tissue to accept a transplant of 4 g/m2 body surface area (BSA) or 0.2 g/kg subject bodyweight;
* Had human immunodeficiency virus (HIV) infection;
* Had prior attempts at immune reconstitution, such as bone marrow transplant or previous thymus transplantation;
* Ventilator support or positive pressure support: Subjects had to be off ventilator or other pressure support such as continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BiPAP) support for 2 weeks prior to enrollment. If the subject was enrolled and was placed back on ventilator or pressure support, the subject had to be able to be weaned off and remain off ventilator or pressure support for 2 weeks. If the subject could not be successfully weaned off ventilator or pressure support, the subject was to be withdrawn from the study.

Additional Inclusion Criteria for Parathyroid Transplant Recipient:

* 2 tests in patient showing: intact parathyroid hormone (PTH) < 5 pg/ml when ionized calcium < 1.1 mmol/L
* All inclusion criteria for thymus transplant must be met
* 2 involved parents

Exclusion for Parathyroid Transplant Recipient:

* Parents do not meet enrollment criteria.
* Parent(s) decline to be parathyroid donor(s).

Parental Parathyroid Donor Inclusion:

* > 18 years old
* Answers all questionnaire items and meets safety screening criteria
* Normal serum calcium
* Normal PTH function
* HLA typing consistent with parentage
* Parent chosen for donation will share HLA-DR allele in thymus donor; if not applicable, then either parent will be selected (if meet all other criteria).
* Must not be on anticoagulation or can come off for donation/transplantation

Parental Parathyroid Donor Exclusion:

* Donor is only living involved parent or caretaker of the recipient
* Hypoparathyroidism - low parathyroid hormone (PTH) in presence of low serum calcium and high serum phosphate
* Hyperparathyroidism (or history of) - elevated PTH in presence of high serum calcium and low serum phosphate
* History of cancer
* Evidence of any of following: HIV-1, HIV-2, HTLV-1, HTLV-2, syphilis, hepatitis B, hepatitis C, West Nile virus, or Trypanosoma Cruzi (Chagas disease)
* Elevated AST, ALT, alkaline phosphatase > 3 times upper limit of normal
* History including receipt of a xenograft or risk factors for SARS, Mad Cow - Disease or smallpox. Note: if parent has Mad Cow Disease risk factors (but not active disease), parent(s) may give permission for transplantation.
* CMV positive urine
* Positive CMV IgM antibodies
* Positive IgM anti-EBV VCA
* On blood thinners and cannot stop for the parathyroid donation
* Elevated PT or PTT (> ULN)
* Platelets < 100,000
* Positive Toxoplasma IgM
* The donor will receive a history and physical; may be excluded based on PI's medical judgment
* Hemoglobin < 9 g/dl
* Infectious lesion on head or neck
* Goiter on ultrasound
* Abnormal fiberoptic laryngoscopy of vocal cords
* Pregnancy
* Positive HSV IgG is not an exclusion; however, post transplantation prophylaxis is needed
* Positive VZV IgG is not an exclusion; however, post transplantation prophylaxis is needed
* Medical concern of otolaryngologist
* Concern by medical psychologist or social worker. Parents are interviewed together and separately regarding following areas: medical history; health habits; substance use; relationships and support; education/work history; mental status/psychological history; readiness for donation.
* Questionnaire (safety screening) responses can lead to exclusion.

Biological Mother of DiGeorge Subject Inclusion Criteria:

* Competent to provide consent
* Willing to provide blood for testing (No other inclusion/exclusion for mother)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-09-02 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Louise Markert, MD, PhD, Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Result] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Result] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Result] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Result] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Result] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Result] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Result] Li B, Li J, Devlin BH, Markert ML. Thymic microenvironment reconstitution after postnatal human thymus transplantation. Clin Immunol. 2011 Sep;140(3):244-59. doi: 10.1016/j.clim.2011.04.004. Epub 2011 Apr 16. PMID 21565561
- [Result] Ciupe SM, Devlin BH, Markert ML, Kepler TB. Quantification of total T-cell receptor diversity by flow cytometry and spectratyping. BMC Immunol. 2013 Aug 6;14:35. doi: 10.1186/1471-2172-14-35. PMID 23914737

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The goal of this study is survival of subjects after cultured thymus tissue implantation (CTTI) regardless of parathyroid co-transplantation. No subject underwent CTTI with parathyroid transplant.
Groups:
- Cultured Thymus Tissue Implantation w Parathyroid Transplant: Cultured Thymus Tissue Implantation (CTTI): Thymus tissue (from unrelated donor), thymus donor and thymus donor's birth mother screened for safety. CTTI done under general anesthesia. Cultured thymus tissue is implanted into quadriceps. Thymus dose at least 4grams/m2 body surface area (0.2 grams/kg body weight) and not >18 grams/m2 body surface area (1.0 grams/kg body weight). At time of CTTI, skin biopsy is obtained to look for preexisting T cells. 2-3 months post-CTTI allograft biopsy done to evaluate for thymopoiesis & graft rejection. At time of biopsy, skin biopsy done to look for T cell clonal populations. Allograft biopsy not done if subject medically unstable. Post-CTTI, subjects followed by immune evaluations, using blood samples.
  Parathyroid Tissue for Transplantation: If both parents meet eligibility criteria, the parent chosen for donation will be the one sharing the parental HLA (Human Leukocyte Antigen)-DR allele that is not in the recipient but is in the thymus donor.
- Cultured Thymus Tissue Implantation: Cultured Thymus Tissue Implantation (CTTI): Thymus tissue (from unrelated donor), thymus donor, and thymus donor's birth mother screened for safety. CTTI is done under general anesthesia. Cultured thymus tissue is implanted into quadriceps. Cultured thymus tissue dose at least 4grams/m2 body surface area (0.2 grams/kg body weight) and not >18 grams/m2 body surface area (1.0 grams/kg body weight). At time of CTTI, skin biopsy obtained to look for preexisting T cells. 2-3 months post-CTTI allograft biopsy done to evaluate for thymopoiesis & graft rejection. At time of biopsy, skin biopsy is done to look for T cell clonal populations. (Allograft biopsy not done if subject medically unstable.) Post-CTTI, subjects followed by immune evaluations, using blood samples.
Period: Overall Study
Arm/Group | Cultured Thymus Tissue Implantation w Parathyroid Transplant | Cultured Thymus Tissue Implantation
Started | 0 | 7
Completed | 0 | 5
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant enrolled is not in efficacy analysis; but is included in the AE analysis. After CTTI, participant was determined to have SCID and not cDGA. Efficacy analysis as reported is on cDGA, without the SCID participant as CTTI cannot lead to T cell development in SCID. AE reporting included all participants.
Groups:
- Cultured Thymus Tissue Implantation: Cultured Thymus Tissue Implantation (CTTI) (previously described as transplantation) is done using allogenic cultured postnatal tissue from unrelated donors.
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 316 (182)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Survival at 1 Year Post-CTTI
Description: Survival at 1 year post CTTI was assessed using the Kaplan Meier Estimated Survival. This mathematical function estimates the survival for a certain length of time.
Time Frame: 1 year post-CTTI
Population: Analysis includes cDGA participants. After CTTI, 1 subject was determined to have SCID and not cDGA. Efficacy analysis as reported is on cDGA, without the SCID subject as CTTI cannot lead to T cell development in SCID. No subjects were enrolled into Arm 1. No subjects received parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Number (95% Confidence Interval); unit: % of participants who survive to 1 year
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 6
% of participants who survive to 1 year | 83 [27.3 to 97.5]

2. Secondary Outcome: Survival at 2 Years Post-CTTI
Description: Survival at 2 years post CTTI was assessed using the Kaplan Meier Estimated Survival. This mathematical function estimates the survival for a certain length of time.
Time Frame: 2 years post-CTTI
Population: as for outcome 1
Measure: Number (97.5% Confidence Interval); unit: % of participants who survive to 2 years
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 6
% of participants who survive to 2 years | 83 [27.3 to 97.5]

3. Secondary Outcome: Immune Reconstitution Efficacy - CD3 T Cells
Description: The development of total CD3 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA participants for the 1 year time point if a CD3 T cell count was performed in the relevant time period. The study was designed to assess survival. No subjects were enrolled into Arm 1. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 4
cells/mm3 | 635 [268 to 1400]

4. Secondary Outcome: Immune Reconstitution Efficacy - CD4 T Cells
Description: The development of total CD4 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA participants for the 1 year time point if a CD4 T cell count was performed in the relevant time period. The study was designed to assess survival. No subjects were enrolled into Arm 1. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 4
cells/mm3 | 499 [224 to 760]

5. Secondary Outcome: Immune Reconstitution Efficacy - CD8 T Cells
Description: The development of total CD8 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA participants for the 1 year time point if a CD8 T cell count was performed in the relevant time period. The study was designed to assess survival. No subjects were enrolled into Arm 1. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 4
cells/mm3 | 116 [47 to 394]

6. Secondary Outcome: Immune Reconstitution Efficacy - Naive CD4 T Cells
Description: The development of naive CD4 T cells at one year as measured using flow cytometry
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA participants for the 1 year time point if a T cell count was performed in the relevant time period. The study was designed to assess survival. No subjects were enrolled into Arm 1. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 4
cells/mm3 | 279 [97 to 476]

7. Secondary Outcome: Immune Reconstitution Efficacy - Naive CD8 T Cells
Description: The development of naïve CD8 T cells at one year as measured using flow cytometry.
Time Frame: 1 year post-CTTI
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 2
cells/mm3 | 214 [124 to 304]

8. Secondary Outcome: Immune Reconstitution Efficacy - Response to Mitogens
Description: The development of a T cell proliferative response to the mitogen phytohemagglutinin.
Time Frame: 1 year post-CTTI
Population: Data were only included on cDGA participants for the 1 year time point if testing was performed in the relevant time period. The study was designed to assess survival. No subjects were enrolled into Arm 1. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Median (Inter-Quartile Range); unit: counts per minute (cpm)
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 4
counts per minute (cpm) | 135016 [84404 to 190928]

9. Secondary Outcome: Thymus Allograft Biopsy
Description: Evidence, on biopsy of the thymus tissue implanted in the recipient muscle, that shows the development of new T cells.
Time Frame: 2 to 3 months post-CTTI
Population: cDGA participants who had a biopsy on the thymus tissue implanted.The study was designed to assess survival. No subjects were enrolled into Arm 1. No subjects received a parathyroid transplant. Therefore, results are reported for Arm 2 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 2
Participants
  Evidence of thymopoiesis | 1
  Evidence of rejection | 0
  Inconclusive for thymopoiesis | 1

ADVERSE EVENTS:
Time Frame: Two years post-CTTI
Description: AE reporting on all participants (cDGA and SCID) who received cultured thymus tissue Implantation (CTTI) (previously described as transplantation). No participants received CTTI with a Parathyroid Transplant.
Arm/Group | Cultured Thymus Tissue Implantation
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation (N=7)
Device related infection (Infections and infestations) | 4 (12)
Pyrexia (General disorders) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (2)
Respiratory tract infection bacterial (Infections and infestations) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count abnormal (Investigations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation (N=7)
Pyrexia (General disorders) | 4 (10)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Pneumonia pseudomonal (Infections and infestations) | 2 (3)
Feeding intolerance (Metabolism and nutrition disorders) | 2 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Catheter site erosion (General disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1)
Viraemia (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Urine electrolytes abnormal (Investigations) | 1 (1)
pH urine increased (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Lactase deficiency (Metabolism and nutrition disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No